CLINICAL TRIAL: NCT02151136
Title: Be Sweet to Toddlers During Needles: RCT of Sucrose Compared to Placebo
Brief Title: Be Sweet to Toddlers: Does Sugar Water Reduce Pain During Blood Work?
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital of Eastern Ontario (Other)
Responsible Party: Principal Investigator, Denise Harrison, Chair in Nursing Care of Children, Youth and Families, Children's Hospital of Eastern Ontario
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11/20E
Record Dates: First submitted 2014-05-28; First posted 2014-05-30 (Estimated); Last update posted 2019-11-07 (Actual); Status verified 2019-11

CONDITIONS: Pain Due to Certain Specified Procedures
Keywords: Sucrose; Pain
MeSH Terms: conditions — Pain | interventions — Sucrose; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 24% sucrose + standard care (Experimental): In addition to standard care (topical anesthetic (Ametop or EMLA) + upright holding + distraction + pacifier, if used), a maximum of 2 ml 24% sucrose will be administered orally in 0.25 ml aliquots 2 minutes prior to the needle insertion, at the time of needle insertion, and repeated at 2 minute intervals until the completion of the procedure
  Interventions: Drug: 24% sucrose; Other: Standard care
- Sterile water + standard care (Placebo Comparator): In addition to standard care (topical anesthetic (Ametop or EMLA) + upright holding + distraction + pacifier, if used), a maximum of 2 ml sterile water will be administered orally in 0.25 ml aliquots 2 minutes prior to the needle insertion, at the time of needle insertion, and repeated at 2 minute intervals until the completion of the procedure
  Interventions: Drug: Sterile water; Other: Standard care

INTERVENTIONS:
Drug: 24% sucrose
  Other Names: TootSweet (NPN 80021492); DandleLion Kisses (NPN 80075819)
  Arms: 24% sucrose + standard care
Drug: Sterile water
  Arms: Sterile water + standard care
Other: Standard care — The current standard of care at the study site is use of topical anesthetic (Ametop or EMLA), upright holding of toddler by parent/caregiver during procedure, use of age appropriate nurse directed distraction, and sucking on a pacifier (if normally used by child)

SUMMARY:
The purpose of this study is to determine whether sugar water (24% sucrose) effectively reduces pain in children ages 12 to 36 months undergoing venipuncture, as measured by pain scores and cry duration.

DETAILED DESCRIPTION:
Background:

Hospitalized children and children undergoing medical care as outpatients are frequently required to undergo needle-related procedures, such as venipuncture for diagnostic purposes and ongoing monitoring (Ellis, Sharp, Newhook, & Cohen, 2004). This procedure causes considerable pain and distress, especially in young children (Humphrey, Boon, van Linden van den Heuvell, & van de Wiel, 1992). Children rate needles as being the most distressing aspect of hospitalization (Kortesluoma & Nikkonen, 2006; Kortesluoma & Nikkonen, 2004), yet they are the most frequently performed skin-breaking procedure for hospitalized children (Cummings, Reid, Finley, McGrath, & Ritchie, 1996; Ellis, et al., 2004; Rennick, McHarg, Dell'Api, Johnston, & Stevens, 2008; Stevens et al., 2011). It is estimated that one-quarter of adults have developed a fear needles, most likely developed during childhood (Taddio et al., 2010; Wright, Yelland, Heathcote, Ng, & Wright, 2009). Being afraid of needles increases the risk of avoidance of needles for immunizations and medical care (Taddio et al., 2009; Wright, et al., 2009). It is therefore crucial that health care researchers and clinicians determine effective pain management strategies for young children, and consistently use such strategies in clinical care.

Rationale:

There is a paucity of evidence to support efficacy and feasibility of pain management strategies during needle-related painful procedures in young children, and uncertainties exist regarding analgesic effects of sweet solutions beyond infancy.

Objectives:

The primary objective of this study is to ascertain whether there is evidence of efficacy of oral 24% sucrose (TootSweet, Natural Product Number (NPN) 80021492; DandleLion Kisses, NPN 80075819) in toddlers (ages 12 to 36 months) compared to placebo (water) during venipuncture, as measured by pain scores and cry duration.

Methods:

A single-centre, phase IV, blinded, two-armed randomized controlled trial (RCT).

Study population: Children aged 12 to 36 months, who are patients in the surgical/medical wards of an urban pediatric tertiary care centre who require venipuncture for the purpose of medically-required venous blood sampling.

Sample size: Data from 140 toddlers; 70 randomized to receive sucrose and 70 randomized to receive water.

Data collection: Enrolled children will be video-recorded during their procedure in order to permit completion of the primary outcome measurement at a later date by researchers blinded to the study solutions who were not part of the data collection process.

Statistical analysis: The primary analysis will consist of a two-way ANOVA with main effects for intervention group and age group. As a secondary analysis, an interaction between intervention and age group will be tested. The primary analysis will be adapted to include adjustment for number of previous hospitalizations and length of current hospitalization and number of venipuncture attempts.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 12-36 months, inclusive
* Children who are patients at CHEO in the 4 East/West or 5 East wards (and overflow unit, when applicable), and the Medical Day Unit
* Children who require venipuncture for the purpose of medically required venous blood sampling
* With the exception of the age criteria, children who are eligible to receive sucrose as per the Sucrose CHEO policy for infants
* Children who have their venipuncture performed by hospital-employed phlebotomists or registered nurses (to ensure standardization of the blood collection procedure)
* Parents/guardians and children must also be able to understand English or French

Exclusion Criteria:

* Children who have received a muscle relaxant, opioid analgesic or sedative in the past 24 hours (to ensure there is no interaction effect of these medications which may impact on toddlers' ability to mount a behavioral response to pain)
* Children who are ineligible to receive sucrose as per the Sucrose CHEO policy
* Children who are already consuming sweet fluids or foods, or if the mother wishes to breast feed during the procedure will also be excluded
* Children with known or suspected fructose intolerance

Ages: 12 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 86 (Actual)
Dates: Start 2015-11; Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Cry duration | Cry time will be measured from the time of needle insertion up to 30 seconds after the end of the venipuncture procedure
  Cry is a valid measure of distress in young children and is an objective and easily measurable parameter.

SECONDARY OUTCOMES:
FLACC (Face, Legs, Arms, Crying, Consolability) | FLACC scores will be completed before and during the procedure and up to one minute after the end of the venipuncture procedure
  The FLACC score is a validated 10-point scale composite pain score.
MBPS (Modified Behavioural Pain Scale) | MBPS scores will be completed before and during the procedure and up to one minute after the end of the venipuncture procedure
  The MBPS is a validated 10-point scale composite pain score.
Child's compliance with intervention | up to one minute
  The child's compliance with the study solution during venipuncture will be recorded by the research personnel on the data collection sheet as a 3-point scale (Fully compliant, Somewhat compliant, Not compliant) and will be scored and documented following completion of the procedure. The research personnel will ask the parent or nurse in attendance, what they consider the child's compliance score was.

CONTACTS AND LOCATIONS:
Overall Officials: Denise Harrison, RN, PhD, Principal Investigator — Children's Hospital of Eastern Ontario
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Ellis JA, Sharp D, Newhook K, Cohen J. Selling comfort: A survey of interventions for needle procedures in a pediatric hospital. Pain Manag Nurs. 2004 Dec;5(4):144-52. doi: 10.1016/j.pmn.2004.09.002. PMID 15616484
- [Background] Humphrey GB, Boon CM, van Linden van den Heuvell GF, van de Wiel HB. The occurrence of high levels of acute behavioral distress in children and adolescents undergoing routine venipunctures. Pediatrics. 1992 Jul;90(1 Pt 1):87-91. PMID 1614786
- [Background] Kortesluoma RL, Nikkonen M. 'The most disgusting ever': children's pain descriptions and views of the purpose of pain. J Child Health Care. 2006 Sep;10(3):213-27. doi: 10.1177/1367493506066482. PMID 16940344
- [Background] Kortesluoma RL, Nikkonen M. 'I had this horrible pain': the sources and causes of pain experiences in 4- to 11-year-old hospitalized children. J Child Health Care. 2004 Sep;8(3):210-31. doi: 10.1177/1367493504045822. PMID 15358886
- [Background] Cummings EA, Reid GJ, Finley AG, McGrath PJ, Ritchie JA. Prevalence and source of pain in pediatric inpatients. Pain. 1996 Nov;68(1):25-31. doi: 10.1016/S0304-3959(96)03163-6. PMID 9251995
- [Background] Stevens BJ, Abbott LK, Yamada J, Harrison D, Stinson J, Taddio A, Barwick M, Latimer M, Scott SD, Rashotte J, Campbell F, Finley GA; CIHR Team in Children's Pain. Epidemiology and management of painful procedures in children in Canadian hospitals. CMAJ. 2011 Apr 19;183(7):E403-10. doi: 10.1503/cmaj.101341. Epub 2011 Apr 4. PMID 21464171
- [Background] Rennick JE, McHarg LF, Dell'Api M, Johnston CC, Stevens B. Developing the Children's Critical Illness Impact Scale: capturing stories from children, parents, and staff. Pediatr Crit Care Med. 2008 May;9(3):252-60. doi: 10.1097/PCC.0b013e31816c70d4. PMID 18446107
- [Background] Taddio A, Appleton M, Bortolussi R, Chambers C, Dubey V, Halperin S, Hanrahan A, Ipp M, Lockett D, MacDonald N, Midmer D, Mousmanis P, Palda V, Pielak K, Riddell RP, Rieder M, Scott J, Shah V. Reducing the pain of childhood vaccination: an evidence-based clinical practice guideline. CMAJ. 2010 Dec 14;182(18):E843-55. doi: 10.1503/cmaj.101720. Epub 2010 Nov 22. No abstract available. PMID 21098062
- [Background] Wright S, Yelland M, Heathcote K, Ng SK, Wright G. Fear of needles--nature and prevalence in general practice. Aust Fam Physician. 2009 Mar;38(3):172-6. PMID 19283260
- [Background] Taddio A, Chambers CT, Halperin SA, Ipp M, Lockett D, Rieder MJ, Shah V. Inadequate pain management during routine childhood immunizations: the nerve of it. Clin Ther. 2009;31 Suppl 2:S152-67. doi: 10.1016/j.clinthera.2009.07.022. PMID 19781434